CLINICAL TRIAL: NCT05525715
Title: A Study of Phase Ⅰb/II to Evaluate the Safety, Efficacy and Pharmacokinetic Characteristics of QY201 Tablet in Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study of QY201 Tablet in Subjects With Moderate to Severe Atopic Dermatitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: E-nitiate Biopharmaceuticals (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QY201-Ⅰ-2
Record Dates: First submitted 2022-08-28; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Phase Ib Cohort 1（2mg QY201 tablets or 2mg QY201 placebo） (Experimental): 8 subjects use 2mg QY201 tablets，2 subject uses 2mg QY201 placebo ，BID，29 days
  Interventions: Drug: 2mg QY201 tablets or 2mg QY201 placebo,BID
- Phase Ib Cohort 2（5mg QY201 tablets or 5mg QY201 placebo） (Experimental): 8 subjects use 5mg QY201 tablets，2 subject uses 5mg QY201 placebo ，BID，29 days
  Interventions: Drug: 5mg QY201 tablets or 5mg QY201 placebo,BID
- Phase Ib Cohort 3（10mg QY201 tablets or 10mg QY201 placebo） (Experimental): 8 subjects use 10mg QY201 tablets，2 subject uses 10mg QY201 placebo，QD，29 days
  Interventions: Drug: 10mg QY201 tablets or 10mg QY201 placebo,QD
- Phase Ib Cohort 4（10mg QY201 tablets or 10mg QY201 placebo） (Experimental): 8 subjects use 10mg QY201 tablets，2 subject uses 10mg QY201 placebo，BID，29 days
  Interventions: Drug: 10mg QY201 tablets or 10mg QY201 placebo,BID
- Phase Ib Cohort 5（15mg QY201 tablets or 15mg QY201 placebo） (Experimental): 8 subjects use 15mg QY201 tablets，2 subject uses 15mg QY201 placebo，BID，29 days
  Interventions: Drug: 15mg QY201 tablets or 15mg QY201 placebo,BID
- Phase Ib Cohort 6（20mg QY201 tablets or 20mg QY201 placebo） (Experimental): 8 subjects use 20mg QY201 tablets，2 subject uses 20mg QY201 placebo，BID，29 days
  Interventions: Drug: 20mg QY201 tablets or 20mg QY201 placebo,BID
- Phase II Cohort1 (5mg QY201 tablets) (Experimental): 50 subjects use 5mg QY201 tablets twice daily for 12 weeks
  Interventions: Drug: 5mg QY201 tablets，BID
- Phase II Cohort2 (10mg QY201 tablets) (Experimental): 50 subjects use 10mg QY201 tablets twice daily for 12 weeks
  Interventions: Drug: 10mg QY201 tablets，BID
- Phase II Cohort3 (20mg QY201 tablets) (Experimental): 50 subjects use 20mg QY201 tablets twice daily for 12 weeks
  Interventions: Drug: 20mg QY201 tablets，BID
- Phase II Cohort4 (QY201 placebo) (Experimental): 50 subjects use QY201 placebo twice daily for 12 weeks
  Interventions: Drug: QY201 placebo，BID

INTERVENTIONS:
Drug: 2mg QY201 tablets or 2mg QY201 placebo,BID — 2mg QY201 tablets or 2mg QY201 placebo,BID
  Arms: Phase Ib Cohort 1（2mg QY201 tablets or 2mg QY201 placebo）
Drug: 5mg QY201 tablets or 5mg QY201 placebo,BID — 5mg QY201 tablets or 5mg QY201 placebo,BID
  Arms: Phase Ib Cohort 2（5mg QY201 tablets or 5mg QY201 placebo）
Drug: 10mg QY201 tablets or 10mg QY201 placebo,QD — 10mg QY201 tablets or 10mg QY201 placebo,QD
  Arms: Phase Ib Cohort 3（10mg QY201 tablets or 10mg QY201 placebo）
Drug: 10mg QY201 tablets or 10mg QY201 placebo,BID — 10mg QY201 tablets or 10mg QY201 placebo,BID
  Arms: Phase Ib Cohort 4（10mg QY201 tablets or 10mg QY201 placebo）
Drug: 15mg QY201 tablets or 15mg QY201 placebo,BID — 15mg QY201 tablets or 15mg QY201 placebo,BID
  Arms: Phase Ib Cohort 5（15mg QY201 tablets or 15mg QY201 placebo）
Drug: 20mg QY201 tablets or 20mg QY201 placebo,BID — 20mg QY201 tablets or 20mg QY201 placebo,BID
  Arms: Phase Ib Cohort 6（20mg QY201 tablets or 20mg QY201 placebo）
Drug: 5mg QY201 tablets，BID — 5mg QY201 tablets，BID
  Arms: Phase II Cohort1 (5mg QY201 tablets)
Drug: 10mg QY201 tablets，BID — 10mg QY201 tablets，BID
  Arms: Phase II Cohort2 (10mg QY201 tablets)
Drug: 20mg QY201 tablets，BID — 20mg QY201 tablets，BID
  Arms: Phase II Cohort3 (20mg QY201 tablets)
Drug: QY201 placebo，BID — QY201placebo，BID
  Arms: Phase II Cohort4 (QY201 placebo)

SUMMARY:
This is a phase Ib/II, randomized, double-blind, placebo-controlled, parallel, multicenter study of a certain phase to evaluate the efficacy, safety, and pharmacokinetic characteristics of QY201 tablet in subjects in moderate to severe atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

1. Having been informed the purpose, nature, methods and possible adverse reactions of the trial, the subjects agreed to be subjects and sign an informed consent form before the start of any research process.
2. Part1（Phase Ⅰb）：Male and female subjects aged 18 to 65 (including 18 and 45).Part2（Phase Ⅱ）：Male and female subjects aged 18 to 75 (including 18 and 45).
3. Atopic dermatitis with a diagnosis confirmed by a dermatologist (according to the Hanifin and Rajka criteria); and also onset of symptoms at least 6 month prior to screening visit.
4. Moderate to severe atopic dermatitis defined by an IGA score ≥ 3，an EASI ≥ 16, an PP-NRS≥4, and an BSA ≥ 10% at the screening and baseline visit.
5. Documented history (within 6 mouths prior to the screening visit) of inadequate or medically inadvisable response to topical corticosteroids (TCS), topical calcineurin inhibitors (TCI), systematic treatment or phototherapy.
6. Twice daily use of an stable-dose, additive-free, bland emollient for at least 7 days prior to Day 1, and continued for the duration of this trial.
7. Communicate well with investigators, understand and abide by requirements of this trial.

Exclusion Criteria:

1. Have evidence of active or latent or inadequately treated infection with mycobacterium tuberculosis (TB) as defined by investigators or specialist physicians according to history, symptoms, signs, laboratory tests, T-SPOT test,and imagings, unless subjects had previously received an adequate course of therapy at least 1 month.
2. History of mental disorders, genetic history of mental disorder, or epilepsy treated by antipsychotics and sedatives.
3. In addition to AD, subjects who have current or recent history of clinically significant severe immunologic/rheumatologic, cardiovascular, hepatic, renal, gastrointestinal, or neurologic disease, or have a history of malignancies with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ that might need systematic hormone therapy or other interventions, may increase the risk defined by investigators.
4. In addition to AD, subjects have other dermatoses that affect the evaluation of trial results, or have a wide range of tattoos, birthmarks, skin scars in the skin lesion area.
5. Have a known immunodeficiency disorder or a first-degree relative with a hereditary immunodeficiency.
6. Subjects who have received or are planning to receive an organ transplant operation and are taking immunosuppressants, such as liver or kidney transplantation.
7. Any of the following abnormalities:

   1. Within 3 months, subjects who have acute myocardial infarction, unstable angina pectoris, coronary artery bypass grafting, or coronary stent implantation prior to Day 1;
   2. Have a history of severe arrhythmias, such as (Grade II type 2 or III ATV block, long QT syndrome, or QTcF abnormalities: >470 ms in men and >480 ms in women);
   3. Decompensated cardiac insufficiency (NYHA Class III or IV);
   4. Other cardiac conditions that required treatment and are ineligible for the study according to the investigator.
8. Infected with various viruses. For Hepatitis B, subjects who are Hepatitis B Surface Antigen (HBsAg) or Hepatitis B Core Antibody (HBcAb) positive, and HBV-DNA positive are not eligible for the study. For hepatitis C, subjects who are HCV antibody positive is excluded. Subjects who are Human Immunodeficiency Viruses antibody or Treponema pallidum antibody positive are also not eligible for the study.
9. Presence of any of the following laboratory abnormalities at the screening visit:

   1. Part 1 (Phase Ⅰb):

      Fasting blood glucose>Upper limit of normal (ULN);Hypertension poorly controlled by medication (Systolic pressure≥150mmHg, Diastolic pressure≥95mmHg);WBC, Neutrophils, Lymphocyte count, Platelet count or Hemoglobin<lower limits of normal (LLN);Serum creatinine>ULN or eGFR<60 mL/min;Total bilirubin, AST or ALT values>ULN;PT or APTT values>ULN;
   2. Part 2 (Phase Ⅱ):

   Fasting blood glucose poorly controlled>10 mmol/L;Hypertension poorly controlled by medication (Systolic pressure≥160mmHg, Diastolic pressure≥100mmHg);WBC<3.0×109/L, Neutrophils<1.5×109/L; Lymphocyte count<0.8×109/L, Platelet count<100.0×109/L and Hemoglobin<100 g/L;Serum creatinine>1.5 times the ULN or eGFR<40 mL/min;Total bilirubin>1.5 times the ULN, AST or ALT values>2 times the ULN;PT or APTT values>1.5 times the ULN.
10. Have a clinical symptomatic infection requiring antimicrobial therapy, such as bacteria, viruses, parasites or fungi during screening.
11. Have a history (single episode) of disseminated herpes zoster or disseminated herpes simplex, or a recurrent (more than one episode ) of localized, dermatomal herpes zoster.
12. Have a history of cerebral hemorrhage or cerebral infarction within 1 years prior to Day 1.
13. Have a history of alcohol or substance abuse within 6 months prior to Day 1.
14. Have a history of hemorrhage (more than 400 mL), such as trauma, blood collection or donation, or have a plan of blood donation during or after the study.
15. Have been treated by JAK inhibitors, such as Ruxolitinib, Tofacitinib, Baricitinib, Filgotinib, Lestaurtinib, Pacritinib, Delgocitinib, Upadacitinib, or Abrocitinib, within 3 months prior to Day 1.
16. Have been treated by biologicals of AD, such as Dupilumab, within 8 weeks or 5 half-live prior to Day 1, whichever is longer.
17. Have received grade 3 or 4 surgery within 8 weeks prior to Day 1.
18. Have been vaccinated with live or attenuated live vaccine within 4 weeks prior to Day 1.
19. Prior to Day 1, have joined any clinical trial of drug within 4 weeks (or 5 half-life periods, depending on the longer one), or any clinical trial of medical apparatus and instruments within 3 months.
20. Have been treated by any long-acting anticoagulant drugs, such as Warfarin, Clopidogrel, or subjects who require continuous anticoagulant therapy, except for Aspirin≤100 mg per day.
21. Have a history of oral immune suppressants (eg, systemic corticosteroids, cyclosporine A [CsA], mycophenolate-mofetil [MMF], interferon-γ [IFN-γ], azathioprine, methotrexate) or Phototherapy (eg, UVB or PUVA) within 4 weeks or within 5 half-lives (if known) prior to Day 1, whichever is longer.
22. Have received topical treatments that could affect atopic dermatitis (eg, corticosteroids (TCS), calcineurin inhibitors (TCI), or PDE-4 inhibitors) within 2 weeks prior to Day 1.
23. Have received strong inhibitors or inducers of CYP3A Hepatic metabolic enzymes.
24. Subjects who are unable to take tablets, allergic to the active ingredient or excipient of the investigational drug.
25. In the opinion of the investigator, subjects have a history of gastrointestinal diseases that will affect the absorption of oral drugs, such as gastrointestinal perforation.
26. Pregnant female subjects, breastfeeding female subjects, or male subjects able to father children and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 6 months after last use of investigational drug.
27. Subjects who are unavoidable to or plan exposure to natural or artificial ultraviolet (UV) radiation which could affect atopic dermatitis in the opinion of the investigator.
28. In the opinion of the investigator, subjects who are not suitable to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (AEs)- Phase Ⅰb | From the first administration to 28 days after the last administration of the study drug
  Number of participants with treatment emergent adverse events (AEs) and change from baseline in vital signs (blood pressure, pulse rate, respiratory rate body temperature), physical examination, ECG parameters, clinical laboratory
Percentage of Participants Achieving >=75% Improvement From Baseline in Eczema Area and Severity Index (EASI75) Response at Week 12- Phase Ⅱ | Week 12
  EASI quantifies severity of AD based on severity of lesion clinical signs and percentage (%) of body surface area (BSA) affected. Severity of clinical signs of AD lesions (erythema, induration/papulation, excoriation and lichenification) were scored separately for each of 4 body regions (head and neck, upper limbs, trunk and lower limbs ) on a 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based on % BSA with AD in body region: 0 (0%), 1 (0 to 9%), 2 (10 to 29%), 3 (30 to 49%), 4 (50 to 69%), 5 (70 to 89%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, with higher scores indicating greater severity of AD.

SECONDARY OUTCOMES:
Pharmacokinetic parameters-Phase Ib | Day1 to Day 30
  Tmax
Pharmacokinetic parameters-Phase Ib | Day1 to Day 30
  Cmax
Pharmacokinetic parameters-Phase Ib | Day1 to Day 30
  t1/2
Pharmacokinetic parameters-Phase Ib | Day1 to Day 30
  AUC0-t
Pharmacokinetic parameters-Phase Ib | Day1 to Day 30
  CL/F
Pharmacokinetic parameters-Phase Ib | Day1 to Day 30
  Vz/F
Percentage of Participants Achieving >=50%/75%/90% Improvement From Baseline in Eczema Area and Severity Index (EASI-50/EASI-75/EASI-90) Response at Week 2 and 4 | Week 2 and 4
  EASI quantifies severity of AD based on severity of lesion clinical signs and percentage (%) of body surface area (BSA) affected. Severity of clinical signs of AD lesions (erythema, induration/papulation, excoriation and lichenification) were scored separately for each of 4 body regions (head and neck, upper limbs, trunk and lower limbs ) on a 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based on % BSA with AD in body region: 0 (0%), 1 (0 to 9%), 2 (10 to 29%), 3 (30 to 49%), 4 (50 to 69%), 5 (70 to 89%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, with higher scores indicating greater severity of AD.
Number of Participants With Treatment Emergent Adverse Events (AEs)- Phase Ⅱ | From the first administration to 28 days after the last administration of the study drug
  Number of participants with treatment emergent adverse events (AEs) and change from baseline in vital signs (blood pressure, pulse rate, respiratory rate body temperature), physical examination, ECG parameters, clinical laboratory

CONTACTS AND LOCATIONS:
Overall Officials: LiMing Wu, Ph.D, M.D, Principal Investigator — Affiliated Hangzhou First People's Hospital of Zhejiang University School of Medicine

IPD SHARING:
Plan to Share IPD: No